CLINICAL TRIAL: NCT01482299
Title: A Phase II Trial of RAD001 (Everolimus) for 2nd Line Treatment After Failure of Fluoropyrimidine Plus Platinum Chemotherapy in Patients With Metastatic or Recurrent Gastric Cancer With pS6 Ser 240/4 Expression
Brief Title: RAD001 in Advanced Gastric Cancer Who Failed Standard First-line Treatment With pS6 Ser 240/4 Expression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Yoon-Koo Kang, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC1104
Record Dates: First submitted 2011-11-03; First posted 2011-11-30 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Stomach Neoplasm
Keywords: pS6 Ser 240/4; RAD001 (everolimus); second-line treatment; advanced gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RAD001 (everolimus) (Experimental)
  Interventions: Drug: RAD001

INTERVENTIONS:
Drug: RAD001 — RAD001 (everolimus) 10 mg daily, orally without interruption.
  1 cycle is equal to 4-week treatment. Treatment will be continued unless disease progression or intolerability.
  Other Names: everolimus

SUMMARY:
This is a phase II study to evaluate RAD001 (Everolimus) in terms of 4-month progression-free survival rate (primary end-point) and response rate, toxicity, overall survival and biomarker assessment (secondary end-points) in patients with metastatic or recurrent gastric cancer with pS6 Ser 240/4 expression.

Eligibility criteria include pathologically proven non-resectable adenocarcinoma of stomach with measurable disease who failed previous first-line palliative chemotherapy including fluoropyrimidine and platinum with high expression of pS6 Ser 240/4.

Oral RAD001 (everolimus) 10mg daily will be administered and the dose will be adjusted according to the observed clinical toxicities. Treatment will be continued until disease progression or patient's intolerability to the study drug.

A study requires 40 assessable subjects to decide whether the proportion of patients who are free from progression at 4 months (16 weeks), P, is less than or equal to 0.1 or greater than or equal to 0.25 with a target error rate of 0.05 and β of 0.2. If the number of responses is 7 or less, the hypothesis that P >= 0.250 is rejected with a target error rate of 0.200 and an actual error rate of 0.182. If the investigators assume that drop-out rate is 10%, total accrual patient will be 45.

DETAILED DESCRIPTION:
Methodology: Prospective, non blinded, open label, single center phase II study

Criteria for evaluation: Assessment of response will be assessed radiologically according to RECIST criteria after completion of the two cycles. Evaluation will be by physical examination, chest X-ray, abdomen-pelvis CT scan Safety criteria: Physical examination, vital signs, performance status, CBC, serum chemistry, NCI CTC V.3.0

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically documented stomach adenocarcinoma including adenocarcinoma of the esophagogastric junction
* non-resectable disease by metastasis or recurrent disease after curative surgical resection (See Appendix A) with uni-dimensionally measurable disease
* failure of 1st line chemotherapy including fluoropyrimidine (capecitabine, S1, or 5-FU,) and platinum (cisplatin or oxaliplatin) in palliative setting; progression during or within 6 months after chemotherapy
* High expression of pS6 Ser 240/4 (proportion of pS6 Ser 240/4 positive cancer cells by immunohistochemistry > 10%)
* Age 20 to 75 years old
* Estimated life expectancy of more than 3 months
* ECOG performance status of 2 or lower
* Adequate bone marrow function
* Adequate kidney function
* Adequate liver function
* Fasting serum cholesterol ≤ 300 mg/dL AND fasting triglyceride ≤ 2.5 X ULN
* No prior radiation therapy to more than 25% of BM
* psychological, familial, sociological or geographical conditions which do not permit medical follow-up and compliance with this study
* Women of childbearing potential must have a negative pregnancy test on admission
* Written informed consent

Exclusion Criteria:

* Other tumor type than adenocarcinoma
* CNS metastases or prior radiation for CNS metastases
* Gastric outlet obstruction or intestinal obstruction
* Evidence of active gastrointestinal bleeding
* Bone lesions as the sole evaluable disease
* Past or concurrent history of neoplasm other than stomach cancer
* Pregnant or lactating women, women of childbearing potential not employing adequate contraception
* Other serious illness or medical conditions
* Concomitant or with a 4-week period administration of any other experimental drug under investigation
* Concomitant chemotherapy, hormonal therapy, or immunotherapy
* Any preexisting medical condition of sufficient severity to prevent full compliance with the study

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
4-month progression-free survival | up to 3years
  Progression-free survival is defined as the time from the first treatment to the onset of progressive disease per RECIST criteria or to the date of death whichever comes first. For patients who do not experience progressive disease or death, the progression-free survival duration will be right censored on the last disease assessment date.

SECONDARY OUTCOMES:
Response rate | Up to 1year
  evaluated with abdominal and pelvic dynamic CT scan every 8 weeks, using RECIST version 1.0
Number of participants with adverse events | Monitoring of adverse events will be contineud for at least 28days following the last dose of study treatment
  Adverse events will be graded according to Common Terminology Criteria for Adverse events version 4.0
Overall survival | Up to 3years
  Overall survival duration is calculated as time from the first treatment to the date of death. For patients who are still alive at the cut-off date for statistical reporting, the overall survival duration will be right censored on the last known alive date.
Biomarker assessment | 24months
  Tumor tissues obtained by tumor tissues can be used for immunohistochemistry(IHC) of pS6 Ser 240/4. In patients who did not receive gastrectomy tumor biopsies will be obtained at screening(before everolimus treatment) and after two cycles of treatment. Scoring of all IHC results is based on the percentage of positive cells. The percentage of positive cells is scored as: 0 (0%); 1 (≤10%); 2 (11-33%); 3 (34-66%); 4 (≥67%).

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Koo Kang, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Songpa-gu, Seoul, South Korea